CLINICAL TRIAL: NCT04815759
Title: Dental Anxiety Among Egyptian Children Pre and Post COVID 19
Brief Title: Dental Anxiety Among Children Pre and Post COVID 19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Other Study IDs: Dental anxiety
Record Dates: First submitted 2021-03-20; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre pandemic
  Interventions: Other: routine dental restorative procedures
- Post pandemic
  Interventions: Other: routine dental restorative procedures

INTERVENTIONS:
Other: routine dental restorative procedures — pulp and restorative therapy

SUMMARY:
Dental fear and anxiety is a significant issue that affects pediatric patients and creates challenges in oral health management. Considering that the coronavirus disease 2019 (COVID-19) pandemic, along with its associated sanitary regime, social distancing measures and nationwide quarantines, could itself induce public fears, including in children, it is of great interest to explore whether this situation and the necessity of reorganizing dental care could potentially affect the emotional state of pediatric patients facing a need for urgent dental intervention

ELIGIBILITY:
Inclusion Criteria:

* parental consent
* no previous dental experience
* medically free children

Exclusion Criteria:

* children with negative behavior according to Frankl Rating Scale
* children require general anesthesia

Ages: 4 Years to 6 Years | Sex: All
Age Groups: Child
Study Population: children with an age range 4-6 years attending the outpatient clinic of the of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Alexandria University
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04-27 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Dental anxiety level | through study completion, an average of 3 months
  Assessment will performed by using Facial image scale (FIS)It consists of 5 faces ranging from very happy to very unhappy.
  At the beginning, the 5 faces have been explained to all children and they were asked to point to the face which best describes how he/she felt at the moment

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt